CLINICAL TRIAL: NCT04210518
Title: Influence of Stroboscopic Vision on Balance in Patients With Chronic Ankle Instability
Brief Title: Balance Training With Stroboscopic Vision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Collaborators: University of Miami (Other)
Responsible Party: Principal Investigator, DAVID CRUZ DÍAZ, Professor, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UJASB
Record Dates: First submitted 2019-12-08; First posted 2019-12-24 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Ankle Inversion Sprain; Proprioceptive Disorders
MeSH Terms: conditions — Somatosensory Disorders

STUDY DESIGN:
Intervention Model Description: This study was a single-blinded randomized controlled trial with two intervention groups consisted in multimodal balance training, multimodal balance training in addition to stroboscopic glasses and control group.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: An independent assessor blinded to the data collection was responsible for the allocation process. A list of the computer-generated number was employed to assign participants to balance training group, balance training with stroboscopic glasses group or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neuromuscular training (Experimental): Neuromuscular training consisting of:
  * Single limb balance task.
  * Balance training on an unstable surface.
  * Hop drills.
  Interventions: Other: Neuromuscular training
- Stroboscopic glasses group (Experimental): This group performed the same neuromuscular training with the addition of stroboscopic glasses during the training performance.
  * Single limb balance task.
  * Balance training on unstable surfaces.
  * Hop drills.
  Interventions: Other: Stroboscopic glasses
- Control group (No Intervention): This group received no intervention

INTERVENTIONS:
Other: Neuromuscular training — This intervention consisted of a supervised multimodal exercise protocol addressing different aspects of balance including static and dynamic tasks on the injured ankle. The training program comprised 6 exercises that were progressively adapted depending on the patient's execution controlled by an expert physiotherapist
  Arms: Neuromuscular training
Other: Stroboscopic glasses — Patients included in this group performed the same protocol described in the balance training group with the addition of the stroboscopic glasses during the intervention.
  Arms: Stroboscopic glasses group

SUMMARY:
Balance training with stroboscopic vision in patients with chronic ankle instability.

DETAILED DESCRIPTION:
This study was a single-blinded randomized controlled trial with two intervention groups consisted in multimodal balance training, multimodal balance training in addition to stroboscopic glasses and control group who received no intervention.

ELIGIBILITY:
Inclusion Criteria:

* a previous episode of ankle sprain in at least 6 months before the beginning of the study
* a score of 25 or less in the Cumberland Ankle Instability Tool
* no history of others musculoskeletal injuries in the lower limbs

Exclusion Criteria:

* an acute ankle sprain within the last six weeks
* Recent lower limb surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-20 (Actual)

PRIMARY OUTCOMES:
Ankle range of motion | From baseline to six weeks.
  Ankle dorsiflexion range of motion was assessed by the weight-bearing lunge test. The patient is positioned in a standing position facing a wall with the involved foot parallel with a tape measure which has been attached to the floor and the opposite leg placed behind in a tandem stance. A forward lunge is performed until the anterior knee tries to make contact with the wall with the heel firmly planted on the ground.
Dynamic balance | From baseline to six weeks.
  Dynamic balance has been measured by a simplified version of the Star Excursion Balance Test where the anterior, posteromedial and posterolateral reach directions were collected for statistical analysis.

SECONDARY OUTCOMES:
Self-reported instability and function | From baseline to six weeks.
  To determine the severity of ankle instability the Cumberland ankle instability tool. This questionnaire is a nine items questionnaire ranged from 0 to 30 (0 related with severe impairment and 30 no subjective instability feeling) and has been reported to be a valid tool with high internal consistency and reliability.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Jaen, Jaén, Spain

IPD SHARING:
Plan to Share IPD: No